CLINICAL TRIAL: NCT02591238
Title: The Protective Effect of Melatonin on Smoke-induced Vascular Injury in Human
Brief Title: Melatonin in Smoke-induced Vascular Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 81470585
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-06

CONDITIONS: Smoking; Vascular System Injuries
Keywords: smoking; melatonin; vascular injury
MeSH Terms: conditions — Smoking; Vascular System Injuries | interventions — Melatonin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-smoker + placebo (Placebo Comparator): non-smoker oral placebo
  Interventions: Other: non-smoker oral placebo
- non-smoker + melatonin (Active Comparator): non-smoker oral melatonin
  Interventions: Drug: non-smoker oral melatonin
- smoker + placebo (Placebo Comparator): smoker oral placebo
  Interventions: Other: smoker oral placebo
- smoker + melatonin (Active Comparator): smoker oral melatonin
  Interventions: Drug: smoker oral melatonin

INTERVENTIONS:
Other: non-smoker oral placebo — Participants oral placebo last 2 weeks.
  Other Names: placebo
  Arms: non-smoker + placebo
Drug: non-smoker oral melatonin — Participants oral melatonin 3 mg/day last 2 weeks.
  Other Names: Melatonin
  Arms: non-smoker + melatonin
Other: smoker oral placebo — Participants oral placebo last 2 weeks.
  Other Names: placebo
  Arms: smoker + placebo
Drug: smoker oral melatonin — Participants oral melatonin 3 mg/day last 2 weeks.
  Other Names: melatonin
  Arms: smoker + melatonin

SUMMARY:
The main purpose of this study was to evaluate the effects of melatonin in the regulation of the vascular injury in smokers through population-based, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Trial title: The protective effect of melatonin on smoke-induced vascular injury in human

Protocol: Investigators recruited eligible Han Chinese participants (aged 25-39) if they had smoking at least 10 cigarettes per day for at least 1 year. Participants excluded if they had undergone cardiovascular disease, or systolic blood pressure above 140 mm Hg, or diastolic blood pressure above 90 mmHg, or psychiatric disorders, or cancer, or pregnant, or lactating, or taking antipsychotic drugs orally during the 2 weeks of the trial. They were randomly divided participants into non-smoking with oral placebo, non-smoking with oral melatonin, smoking with oral placebo, and smoking with oral melatonin. They are oral melatonin 3 mg/day or placebo for 2 weeks. Blood samples (about 3 milliliter) were taken at baseline and after 2 weeks of treatment. Through a series hospital clinical laboratory and related ELISA kits to detect endothelial cell injury in serum markers platelet endothelial cell adhesion molecule-1 (PECAM-1/CD31)， intercellular adhesion molecule-1 (ICAM - 1), vascular cell adhesion molecule-1 (VCAM 1), endothelin-1 (ET-1), endothelial nitric oxide synthase (eNOS), nuclear erythroid 2-related factor 2 (Nrf - 2), NAD(P)H quinone oxidoreductase-1 (NQO-1), catalytic glutamate cysteine ligase (GCLC), heme oxygenase-1 (HO-1), free fatty acid (FFA), total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL), hypersensitive c-reactive protein (hsCRP), fibrinogen (Fbg), and free fatty acids (FFA), through the above vascular endothelial damage index analysis whether melatonin have protective effect against smoke-induced vascular injury. All participants and study investigators were unaware of treatment allocation throughout the trial. This trial is approved by the Ethical Committee of Peking Union Medical College Hospital (No JS-863). All participants completed a questionnaire and signed an informed consent document. Otherwise, they will get appropriate economic compensation. To achieve treatment concealment, melatonin and placebo in appearance and package were identically. Trial associates monitored compliance with the masking procedure throughout the trial. All participants and study investigators were unaware of treatment allocation throughout the study. The randomization codes remained sealed until after data collection and cleaning, and completion of a masked analysis. The study team monitored and classified protocol deviations. Investigators summarized baseline clinical and demographic characteristics with descriptive statistics and then determined by the Univariate Analysis of Variance. All the data analyses were done using statistical software SPSS 20.0.

Expected results: Compared with smoker oral placebo, melatonin 3 mg/day may be alleviate smoke-induced vascular injury.

Consent document: The potential risk, research as a treatment drug of melatonin may delay the metabolism of antipsychotic antipsychotic drug, so when investigators recruit psychiatric disorders or taking antipsychotic drugs orally during the 2 weeks of the trial should exclusion. As a Health care medicine. Melatonin is not suitable for children, so investigators selected recruiting participants under the age of 25 to 39.

The measure to minimize the risk, fully inform the participants and their families the trial's advantages, disadvantages and desired effect. All participants totally agree with the subjects. In this process, at least three or more effective way to get contact with the medical staff or doctor and ensure that those unexpected accident should deserve effective tackle. Examination for every participant before start of the trial to guarantee they comply with the criterion. Our research involves the application of melatonin is through the china food and drug administration (CFDA) approved to ensure its safety (include its chemical composition, structure, content parameters, main raw material and appropriate crowd). All staff is qualified medical professionals to guarantee the safety of all participants.

The potential risks or discomfort, or inconvenience, or benefits for participants: So far, effective of melatonin in human include regulating sleep, anti-tumor, immune regulation, regulating of inflammation and immune and regulating blood lipid metabolism is confirmed. Adverse reactions is slow the delay of antipsychotic drug metabolism (so nearly one month ago and during period of the trial participants should not taking antipsychotic drugs) during the trial. The basic principle during the trial is ensure safety of participants.

The relevant content consultation: Everyone have the right to consultation the research content through telephone: +86 01069152500 (principal investigator) and +86 01069155817(Ethics committee).

The rights of withdrew from the trial: Participate in the trial is completely voluntary. If for any reason, participants not willing to participate in, or do not wish to continue to participate in this trial, will not affect the rights and interests of participants. In addition, participants have the right to withdraw this trial at any time. If participants do not according to the doctor instructions, or for the sake of your health and benefits, the doctor or the researchers may also require participants to quit the trial.

The compensation of research: If the participants have any unexpected accident relation with the trial, the compensation and responsibility will be provided by Peking union medical college hospital.

Privacy protection: The privacy of every participant will be protected. The results of the trial in academic publications will not leak any information to identify your personal identity. Peking union medical college hospital will save everybody's data and guarantee not leak without authorization.

Investigators declare no competing interests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers：must above 10 cigarettes per day, at least 1 year
* Healthy non-smokers

Exclusion Criteria:

* Cardiovascular disease
* Systolic blood pressure above 140 mm Hg
* Diastolic blood pressure above 90 mmHg
* Psychiatric disorders
* Cancer
* Pregnant
* Lactating
* Taking antipsychotic drugs orally during the 2 weeks of the trial

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Changwei Liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- PekingUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The cycle of the experiment is long, and it is a part of the experiment.

REFERENCES:
- [Result] Yang GH, Li YC, Wang ZQ, Liu B, Ye W, Ni L, Zeng R, Miao SY, Wang LF, Liu CW. Protective effect of melatonin on cigarette smoke-induced restenosis in rat carotid arteries after balloon injury. J Pineal Res. 2014 Nov;57(4):451-8. doi: 10.1111/jpi.12185. Epub 2014 Oct 6. PMID 25251422
- [Result] Rodella LF, Filippini F, Bonomini F, Bresciani R, Reiter RJ, Rezzani R. Beneficial effects of melatonin on nicotine-induced vasculopathy. J Pineal Res. 2010 Mar;48(2):126-32. doi: 10.1111/j.1600-079X.2009.00735.x. Epub 2009 Dec 30. PMID 20050989
- [Result] Hardeland R, Tan DX, Reiter RJ. Kynuramines, metabolites of melatonin and other indoles: the resurrection of an almost forgotten class of biogenic amines. J Pineal Res. 2009 Sep;47(2):109-126. doi: 10.1111/j.1600-079X.2009.00701.x. Epub 2009 Jul 1. PMID 19573038
- [Result] Hautamaki RD, Kobayashi DK, Senior RM, Shapiro SD. Requirement for macrophage elastase for cigarette smoke-induced emphysema in mice. Science. 1997 Sep 26;277(5334):2002-4. doi: 10.1126/science.277.5334.2002. PMID 9302297
- [Result] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Result] Teo KK, Ounpuu S, Hawken S, Pandey MR, Valentin V, Hunt D, Diaz R, Rashed W, Freeman R, Jiang L, Zhang X, Yusuf S; INTERHEART Study Investigators. Tobacco use and risk of myocardial infarction in 52 countries in the INTERHEART study: a case-control study. Lancet. 2006 Aug 19;368(9536):647-58. doi: 10.1016/S0140-6736(06)69249-0. PMID 16920470
- [Result] Pirie K, Peto R, Reeves GK, Green J, Beral V; Million Women Study Collaborators. The 21st century hazards of smoking and benefits of stopping: a prospective study of one million women in the UK. Lancet. 2013 Jan 12;381(9861):133-41. doi: 10.1016/S0140-6736(12)61720-6. Epub 2012 Oct 27. PMID 23107252
- [Result] Opie LH. The metabolic vicious cycle in heart failure. Lancet. 2004 Nov 13-19;364(9447):1733-4. doi: 10.1016/S0140-6736(04)17412-6. No abstract available. PMID 15541431
- [Result] Bonita R, Magnusson R, Bovet P, Zhao D, Malta DC, Geneau R, Suh I, Thankappan KR, McKee M, Hospedales J, de Courten M, Capewell S, Beaglehole R; Lancet NCD Action Group. Country actions to meet UN commitments on non-communicable diseases: a stepwise approach. Lancet. 2013 Feb 16;381(9866):575-84. doi: 10.1016/S0140-6736(12)61993-X. Epub 2013 Feb 12. PMID 23410607
- [Result] Tan DX, Manchester LC, Reiter RJ, Plummer BF, Hardies LJ, Weintraub ST, Vijayalaxmi, Shepherd AM. A novel melatonin metabolite, cyclic 3-hydroxymelatonin: a biomarker of in vivo hydroxyl radical generation. Biochem Biophys Res Commun. 1998 Dec 30;253(3):614-20. doi: 10.1006/bbrc.1998.9826. PMID 9918777
- [Result] Reiter RJ, Tan DX, Galano A. Melatonin: exceeding expectations. Physiology (Bethesda). 2014 Sep;29(5):325-33. doi: 10.1152/physiol.00011.2014. PMID 25180262
- [Result] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Result] Tan DX, Hardeland R, Manchester LC, Galano A, Reiter RJ. Cyclic-3-hydroxymelatonin (C3HOM), a potent antioxidant, scavenges free radicals and suppresses oxidative reactions. Curr Med Chem. 2014;21(13):1557-65. doi: 10.2174/0929867321666131129113146. PMID 24304286
- [Result] Reiter RJ. Melatonin: Lowering the High Price of Free Radicals. News Physiol Sci. 2000 Oct;15:246-250. doi: 10.1152/physiologyonline.2000.15.5.246. PMID 11390919
- [Result] Rostron BL, Chang CM, Pechacek TF. Estimation of cigarette smoking-attributable morbidity in the United States. JAMA Intern Med. 2014 Dec;174(12):1922-8. doi: 10.1001/jamainternmed.2014.5219. PMID 25317719
- [Result] Bernhard D, Pfister G, Huck CW, Kind M, Salvenmoser W, Bonn GK, Wick G. Disruption of vascular endothelial homeostasis by tobacco smoke: impact on atherosclerosis. FASEB J. 2003 Dec;17(15):2302-4. doi: 10.1096/fj.03-0312fje. Epub 2003 Oct 2. PMID 14525940
- [Result] Pope CA 3rd, Burnett RT, Krewski D, Jerrett M, Shi Y, Calle EE, Thun MJ. Cardiovascular mortality and exposure to airborne fine particulate matter and cigarette smoke: shape of the exposure-response relationship. Circulation. 2009 Sep 15;120(11):941-8. doi: 10.1161/CIRCULATIONAHA.109.857888. Epub 2009 Aug 31. PMID 19720932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Time: Jun 10,2015 -Jun 24,2015. Address: factory clinic of Heilongjiang Airports Managements Group Co., Ltd and village clinic of Xinfa village Daoli district, Haerbin city, Heilongjiang province, China. Medical staff: 3 Registered medical practitioner and 4 registered nurse.
Pre-assignment Details: First in included 96 participants of both genders, 28 participants excluded (refused to randomly assigned n=9, not meeting inclusion criteria n=9, time improper n=8, unknown n=2). 5 participants withdraw during the trial (pregnant n=1, influenza n=1, personal circumstance n=2, unknown reason n=1).
Groups:
- IV Non-smoker + Placebo: non-smoker oral placebo
  non-smoker oral placebo: Participants oral placebo last 2 weeks.
- III Non-smoker + Melatonin: non-smoker oral melatonin
  non-smoker oral melatonin: Participants oral melatonin 3 mg/day last 2 weeks.
- II Smoker + Placebo: smoker oral placebo
  smoker oral placebo: Participants oral placebo last 2 weeks.
- I Smoker + Melatonin: smoker oral melatonin
  smoker oral melatonin: Participants oral melatonin 3 mg/day last 2 weeks.
Period: Overall Study
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Started | 16 | 17 | 17 | 18
Completed | 15 | 16 | 17 | 15
Not Completed | 1 | 1 | 0 | 3
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — influenza | 0 | 0 | 0 | 1
Not completed — personal circumstances | 0 | 0 | 0 | 1
Not completed — personal circumstances | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: According to the requirements of the randomized controlled trials and statistical methods to determine a total of 63 participants, and signed the informed consent.
Groups:
- IVnon-smoker + Placebo: non-smoker oral placebo
  non-smoker oral placebo: Participants oral placebo last 2 weeks.
- IIInon-smoker + Melatonin: non-smoker oral melatonin
  non-smoker oral melatonin: Participants oral melatonin 3 mg/day last 2 weeks.
- IIsmoker + Placebo: smoker oral placebo
  smoker oral placebo: Participants oral placebo last 2 weeks.
- Ismoker + Melatonin: smoker oral melatonin
  smoker oral melatonin: Participants oral melatonin 3 mg/day last 2 weeks.
- Total: Total of all reporting groups
Arm/Group | IVnon-smoker + Placebo | IIInon-smoker + Melatonin | IIsmoker + Placebo | Ismoker + Melatonin | Total
Number analyzed (Participants) | 15 | 16 | 17 | 15 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (3.4) | 34.6 (3.8) | 31.7 (3.4) | 31.7 (2.8) | 33.37 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 14 | 13 | 46
  Male | 6 | 6 | 3 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of Fbg.
Time Frame: Three months
Population: Bellow concentration data of Fbg was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
g/L | 2.76 (0.34) | 2.38 (0.43) | 2.89 (0.58) | 2.49 (0.54)

2. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of Glu.
Time Frame: Three months.
Population: Bellow concentration data of Glu was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
mmol/L | 4.4 (1.36) | 4.24 (1.3) | 5.02 (1.26) | 4.79 (1.05)

3. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of FFA.
Time Frame: Three months.
Population: Below concentration data of FFA was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
umol/L | 389 (121) | 382 (49) | 499 (84) | 425 (64)

4. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of TC.
Time Frame: Three months.
Population: Bellow concentration data of TC was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
mmol/L | 4.51 (1.04) | 4.5 (0.95) | 4.74 (0.8) | 4.45 (0.65)

5. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of TG.
Time Frame: Three months.
Population: Bellow concentration data of TG was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
mmol/L | 1.21 (0.55) | 1.23 (0.6) | 1.42 (0.74) | 1.41 (0.51)

6. Primary Outcome: Smoke-induced Vascular Injury and Melatonin's Effect in This Process Assessed by the Concentration of LDL-C.
Time Frame: Three months.
Population: Bellow concentration data of LDL-C was after treatment with oral melatonin 2 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IV Non-smoker + Placebo | III Non-smoker + Melatonin | II Smoker + Placebo | I Smoker + Melatonin
Number analyzed (Participants) | 15 | 16 | 17 | 15
mmol/L | 1.85 (0.54) | 1.95 (0.52) | 2.2 (0.75) | 2.19 (0.47)

ADVERSE EVENTS:
Time Frame: Any adverse reaction symptoms of all participants were observed for three months.
Description: All participants did not have any adverse reactions during the three month period.
Arm/Group | Non-smoker + Placebo | Non-smoker + Melatonin | Smoker + Placebo | Smoker + Melatonin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/17 | 0/15

LIMITATIONS AND CAVEATS:
Limitations. First, the dose-dependent manner of melatonin should be considered. Second, the duration of smoke exposure and melatonin administration time should be prolonged. Lastly,the levels of melatonin at different time points should be examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes